CLINICAL TRIAL: NCT03694613
Title: A Pilot Study to Evaluate the Utility of Placental/Umbilical Cord Blood (PUCB) in Early Onset Neonatal Sepsis (EONS) in Very Low Birth Weight Infants
Brief Title: Utility of Placental/Umbilical Cord Blood in Early Onset Neonatal Sepsis in Very Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-0165
Record Dates: First submitted 2018-09-28; First posted 2018-10-03 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2020-11

CONDITIONS: Preterm Infant; Early-Onset Neonatal Sepsis; Umbilical Cord
Keywords: Preterm Infant; Early-Onset Neonatal Sepsis; Umbilical Cord; Complete Cell Count; Placenta; Blood Culture
MeSH Terms: conditions — Premature Birth; Neonatal Sepsis

STUDY DESIGN:
Masking Description: Clinical team (care provider) will be blinded to the Placental/Umbilical Cord Blood sepsis evaluation results
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placental/Umbilical Cord Blood sample (Other): Placental/Umbilical Cord Blood sample will be collected after delivery from every participant.
  Interventions: Other: Placental/Umbilical Cord Blood sample

INTERVENTIONS:
Other: Placental/Umbilical Cord Blood sample — After infant is delivered, placenta along with clamped umbilical cord Blood will be obtained from the ObGyn team. One umbilical clamp will be placed at the umbilical end, and the other clamp will be placed on the placental end of the umbilical cord. Then the umbilical cord will be cut between the clamps. The umbilical cord will be cleaned three times with 2% chlorhexidine, plus 70% isopropyl alcohol under sterile conditions (sterile gloves). Cord blood samples will be collected using vacutainer blood collecting system with a sterile 22-gauge needle. We will collect 3 - 4 ml of blood.

SUMMARY:
This study evaluates the utility of placental/umbilical cord blood (PUCB) to perform the baseline workup testing for EONS in Very Low Birth Weight Infants: CBC (Complete Blood Count) with differential, Immature/Total ratio (I/T ratio), and blood culture along with CRP and IL-6 levels. A cohort (63 subjects) of preterm infants will be recruited. All the participants will be evaluated for sepsis using placental/umbilical cord blood (PUCB) and subject blood sample during the first 12 hours of life (after birth).

DETAILED DESCRIPTION:
Early Onset Neonatal Sepsis (EONS) is common in preterm infants, and it is associated with high morbidity and mortality, especially if not diagnosed early. Currently the baseline workup is done using blood samples from the infant to perform Blood culture, CBC, I/T ratio. These tests have shown to have low sensitivity and specificity to diagnosis EONS.

PUCB can be another safe source of blood which is useful, painless and simple to collect. As CBC, I/T ratio and blood culture may not be enough to diagnose EONS we will add IL-6 and CRP which will increase sensitivity and specificity to diagnose EONS in preterm infants without collecting blood from the infants.

This study may be a step to decrease iatrogenic blood loss to diagnose EONS. The primary outcome of the current research will be to find out the utility of PUCB in diagnosing EOS in preterm infants (<30 weeks and <1250 grams birth weight). Using PUCB can increase the accuracy to diagnose Sepsis in Preterm infants, and it will also conserve blood in the extremely premature infants while reducing hemodynamic instability due to acute blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Infants <34 weeks' gestational

Exclusion Criteria:

* Known congenital or chromosomal anomalies
* Congenital heart disease (other than Patent Ductus Arteriosus, Patent Foramen Ovale or Atrial Septum Defect)
* Vaginal bleeding at admission

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sergio M Lerma Narvaez, Principal Investigator — UTMB, Galveston
Locations (1):
- Sergio Mauricio Lerma Narvaez, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qazi SA, Stoll BJ. Neonatal sepsis: a major global public health challenge. Pediatr Infect Dis J. 2009 Jan;28(1 Suppl):S1-2. doi: 10.1097/INF.0b013e31819587a9. No abstract available. PMID 19106756
- [Background] Brown DR, Kutler D, Rai B, Chan T, Cohen M. Bacterial concentration and blood volume required for a positive blood culture. J Perinatol. 1995 Mar-Apr;15(2):157-9. PMID 7595778
- [Background] Hornik CP, Benjamin DK, Becker KC, Benjamin DK Jr, Li J, Clark RH, Cohen-Wolkowiez M, Smith PB. Use of the complete blood cell count in early-onset neonatal sepsis. Pediatr Infect Dis J. 2012 Aug;31(8):799-802. doi: 10.1097/INF.0b013e318256905c. PMID 22531231
- [Background] Malik A, Hui CP, Pennie RA, Kirpalani H. Beyond the complete blood cell count and C-reactive protein: a systematic review of modern diagnostic tests for neonatal sepsis. Arch Pediatr Adolesc Med. 2003 Jun;157(6):511-6. doi: 10.1001/archpedi.157.6.511. PMID 12796229
- [Background] Ng PC. Diagnostic markers of infection in neonates. Arch Dis Child Fetal Neonatal Ed. 2004 May;89(3):F229-35. doi: 10.1136/adc.2002.023838. PMID 15102726
- [Background] Laborada G, Rego M, Jain A, Guliano M, Stavola J, Ballabh P, Krauss AN, Auld PA, Nesin M. Diagnostic value of cytokines and C-reactive protein in the first 24 hours of neonatal sepsis. Am J Perinatol. 2003 Nov;20(8):491-501. doi: 10.1055/s-2003-45382. PMID 14703598
- [Background] Christensen RD, Lambert DK, Baer VL, Montgomery DP, Barney CK, Coulter DM, Ilstrup S, Bennett ST. Postponing or eliminating red blood cell transfusions of very low birth weight neonates by obtaining all baseline laboratory blood tests from otherwise discarded fetal blood in the placenta. Transfusion. 2011 Feb;51(2):253-8. doi: 10.1111/j.1537-2995.2010.02827.x. Epub 2010 Aug 16. PMID 20723166
- [Background] Meena J, Charles MV, Ali A, Ramakrishnan S, Gosh S, Seetha KS. Utility of cord blood culture in early onset neonatal sepsis. Australas Med J. 2015 Aug 31;8(8):263-7. doi: 10.4066/AMJ.2015.2460. eCollection 2015. PMID 26392823
- [Background] Beeram MR, Loughran C, Cipriani C, Govande V. Utilization of umbilical cord blood for the evaluation of group B streptococcal sepsis screening. Clin Pediatr (Phila). 2012 May;51(5):447-53. doi: 10.1177/0009922811431882. Epub 2011 Dec 22. PMID 22199177
- [Background] Joram N, Boscher C, Denizot S, Loubersac V, Winer N, Roze JC, Gras-Le Guen C. Umbilical cord blood procalcitonin and C reactive protein concentrations as markers for early diagnosis of very early onset neonatal infection. Arch Dis Child Fetal Neonatal Ed. 2006 Jan;91(1):F65-6. doi: 10.1136/adc.2005.074245. PMID 16371391
- [Background] Baer VL, Lambert DK, Carroll PD, Gerday E, Christensen RD. Using umbilical cord blood for the initial blood tests of VLBW neonates results in higher hemoglobin and fewer RBC transfusions. J Perinatol. 2013 May;33(5):363-5. doi: 10.1038/jp.2012.127. Epub 2012 Oct 4. PMID 23047426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the Neonatal Intensive Care of the University of Texas Medical Branch, Galveston, Texas.
Pre-assignment Details: We included 65 PI <34 weeks, who were screened for EOS and admitted to the NICU (June 2019 to June 2020). Infants with known lethal chromosomal or congenital anomalies were excluded.
Groups:
- Placental/Umbilical Cord Blood Samples: Study Group: Placental/Umbilical Cord Blood sample will be collected after delivery from every participant recruited.
  Placental/Umbilical Cord Blood sample: After an infant is delivered, placenta along with clamped umbilical cord Blood will be obtained from the ObGyn team. One umbilical clamp will be placed at the umbilical end, and the other clamp will be placed on the placental end of the umbilical cord. Then the umbilical cord will be cut between the clamps. The umbilical cord will be cleaned three times with 2% chlorhexidine, plus 70% isopropyl alcohol under sterile conditions (sterile gloves). Cord blood samples will be collected using a vacutainer blood collecting system with a sterile 22-gauge needle. We will collect 3 - 4 ml of blood.
Period: Overall Study
Arm/Group | Placental/Umbilical Cord Blood Samples
Started | 65
Completed | 65 (65 samples were collected and analyzed. at least 3 ml were collected.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: We recruited 65 subjects (41% female) in the study from June 2019 To June 2020. Gestational age was 32.15 + 2.21 weeks and birth weight 1853 + 519 grams.
Groups:
- Placental/Umbilical Cord Blood Sample: Placental/Umbilical Cord Blood sample will be collected after delivery from every participant.
  Plancental/Umbilical Cord Blood sample: After infant is delivered, placenta along with clamped umbilical cord Blood will be obtained from the ObGyn team. One umbilical clamp will be placed at the umbilical end, and the other clamp will be placed on the placental end of the umbilical cord. Then the umbilical cord will be cut between the clamps. The umbilical cord will be cleaned three times with 2% chlorhexidine, plus 70% isopropyl alcohol under sterile conditions (sterile gloves). Cord blood samples will be collected using vacutainer blood collecting system with a sterile 22-gauge needle. We will collect 3 - 4 ml of blood.
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 32.15 (2.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 41
  More than one race | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65
Birth weight [Mean (Standard Deviation); unit: grams] | 1853 (519)

OUTCOME MEASURES:

1. Primary Outcome: White Blood Cell Count (WBC) (1)
Description: Normal Range approximately 6,000 - 30,000 cell/mm3.
Time Frame: Completed during the first 30 minutes after birth. This sample is going to be taken from the discarded Placental/umbilical blood cord.
Measure: Mean (Standard Deviation); unit: ratio of cells/mm3
Groups:
- Placental/Umbilical Cord Blood Sample: Study Group: Placental/Umbilical Cord Blood sample will be collected after delivery from every participant recruited.
  Plancental/Umbilical Cord Blood sample: After infant is delivered, placenta along with clamped umbilical cord Blood will be obtained from the ObGyn team. One umbilical clamp will be placed at the umbilical end, and the other clamp will be placed on the placental end of the umbilical cord. Then the umbilical cord will be cut between the clamps. The umbilical cord will be cleaned three times with 2% chlorhexidine, plus 70% isopropyl alcohol under sterile conditions (sterile gloves). Cord blood samples will be collected using vacutainer blood collecting system with a sterile 22-gauge needle. We will collect 3 - 4 ml of blood.
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
ratio of cells/mm3 | 8257 (2966)

2. Primary Outcome: White Blood Cell Count (WBC) (1) INFANT BLOOD
Description: Normal Range: 6.000 - 30.000 cell/mm3.
Time Frame: Completed during the first 6 hours after birth. This sample is going to be taken directly from the participant.
Population: Infant blood taken from 65 subjects after birth
Measure: Mean (Standard Deviation); unit: ratio of cells/mm3
Groups:
- WBC- INFANT BLOOD: Blood was taken from all 65 Infants after birth
Arm/Group | WBC- INFANT BLOOD
Number analyzed (Participants) | 65
ratio of cells/mm3 | 7055 (12400)

3. Primary Outcome: I/T Ratio (Immature/Total Immature Neutrophil).I/T Ratio Was Calculated by Dividing Immature White Cell Count Total White Cell Count
Description: Normal Range of I/T ratio: <0.2.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio of Immatures/Total neutrophils
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
Ratio of Immatures/Total neutrophils | 0.09 (0.13)

4. Primary Outcome: I/T Ratio (Immature/Total Immature Neutrophil Ratio) INFANT BLOOD
Description: Normal Range: <0.2
Time Frame: Completed during the first 12 hours after birth. This sample is going to be taken directly from the participant.
Measure: Mean (Standard Deviation); unit: Immatures/Total neutrophils ratio
Groups:
- I/T Ratio. INFANT BLOOD: Blood took from infant
Arm/Group | I/T Ratio. INFANT BLOOD
Number analyzed (Participants) | 65
Immatures/Total neutrophils ratio | 0.12 (0.13)

5. Primary Outcome: CRP (C-Reactive Protein)(1)
Description: Normal Range: < 10,000 ng/mL
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
ng/mL | 413 (1229)

6. Primary Outcome: CRP (C-Reactive Protein)(2) INFANT BLOOD
Description: Normal Range: <10.000ng/mL
Time Frame: Completed during the first 6 hours after birth. This sample was taken directly from the participant.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- CRP- INFANT BLOOD: Blood took from infant
Arm/Group | CRP- INFANT BLOOD
Number analyzed (Participants) | 65
ng/mL | 785 (1846)

7. Primary Outcome: IL-6 (1)
Description: Normal Range: 0-10.2 pg/ml
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
ng/mL
  PUCB | 61.45 (392.7)
  INFANT BLOOD | 45.36 (182.3)

8. Primary Outcome: IL-6 (Interleukin-6) INFANTS BLOOD
Description: Normal Range: <100 pg/mL
Time Frame: Completed during the first 6hours after birth. This sample is going to be taken directly from the participant.
Population: Blood was taken from all 65 Infants from placenta and from baby 6 hours after birth
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- IL-6 - INFANT BLOOD: Blood was taken from all 65 Infants from placenta and from baby 6 hours after birth
Arm/Group | IL-6 - INFANT BLOOD
Number analyzed (Participants) | 65
pg/mL | 45.36 (182.3)

9. Primary Outcome: Procalcitonin PUBC
Description: Blood was taken from PUBC after delivery
Time Frame: Within 30 minutes after delivery
Population: PUBC from all 65 subjects recruited
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Procalcitonin - PUBC: Blood was taken from PUCB
Arm/Group | Procalcitonin - PUBC
Number analyzed (Participants) | 65
pg/mL | 185.9 (374)

10. Primary Outcome: Procalcitonin Level Was Measured in the Blood From Placenta and From the Baby Within 6 Hours After Birth
Description: Procalcitonin levels
Time Frame: Procalcitonin Level was measured in the blood from placenta and in Infant's Blood (within 6 hours)
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Procalcitonin - Infant's Blood: Blood was taken from the Infant's Blood
Arm/Group | Procalcitonin - Infant's Blood
Number analyzed (Participants) | 65
pg/mL | 131.4 (411.7)

11. Primary Outcome: Number of Participants With Negative Blood Culture From Blood Drawn From Placenta and From Baby Within 6 Hours After Birth
Description: Normal Range: Blood Culture Negative
Time Frame: Blood sample drawn from placenta and from baby within 6 hours after birth.
Population: 65 out of 65 subjects were reported to have NEGATIVE blood cultures
Measure: Count of Participants; unit: Participants
Arm/Group | Placental/Umbilical Cord Blood Sample
Number analyzed (Participants) | 65
Participants | 65

12. Primary Outcome: Presepsin- PUBC
Description: Presepsin level was measured in the blood drawn from placenta and from the baby within 6 hours after birth
Time Frame: First 30 min after birth
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PRESEPSIN- PUCB: Blood took from PUCB
Arm/Group | PRESEPSIN- PUCB
Number analyzed (Participants) | 65
ng/mL | 4.6 (1.6)

13. Primary Outcome: Presepsin-Infant's Blood
Description: Levels of presepsin
Time Frame: First 30 min after birth
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- PRESEPSIN- INFANTS BLOOD: Blood took from INFANTS BLOOD
Arm/Group | PRESEPSIN- INFANTS BLOOD
Number analyzed (Participants) | 65
ng/mL | 5.3 (2)

14. Primary Outcome: Number of Participants With a Negative Blood Culture
Description: Blood is taken from infants after birth
Time Frame: first 2 hours after birth
Population: A negative blood culture indicates no infection
Measure: Count of Participants; unit: Participants
Groups:
- Number of Infant's Blood Cultures: Blood is taken from infants after birth,
Arm/Group | Number of Infant's Blood Cultures
Number analyzed (Participants) | 65
Participants | 65

ADVERSE EVENTS:
Time Frame: 12 months
Description: No reported
Arm/Group | Placental/Umbilical Cord Blood Sample
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03694613/Prot_SAP_000.pdf